CLINICAL TRIAL: NCT04827173
Title: Transcutaneous Electrical Nerve Inhibition Using Medium-frequency Alternating Current
Acronym: tMFAEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: f/2021/013
Record Dates: First submitted 2021-03-05; First posted 2021-04-01 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-01

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental)
  Interventions: Procedure: transcutaneous medium-frequency alternating current

INTERVENTIONS:
Procedure: transcutaneous medium-frequency alternating current — Patients receive nerve block of right forearm through transcutaneous medium-frequency alternating current

SUMMARY:
Patients suffering from neurological disorders often exhibit unwanted sensorimotor activities e.g. spasticity, hypersensitisation, hyper- and dystonia and motor disabilities. Currently, several therapeutic interventions are developed and implemented to overcome these unwanted activities e.g. transcutaneous electrical stimulation (TES), oral medication, botulinum neurotoxin injections, local anaesthetics, rehabilitation robotic training and surgery. However, these therapies offer varying results. Compared to analgesic drugs, TES is associated with fewer side effects and has therefore become a popular therapeutic strategy to treat these unwanted sensorimotor activities. To enable this TES strategy, surface electrodes are attached to the skin overlying the site of pain. Next, a low-frequency electrical current (LFC; 1-100 Hz) is applied. However, this low-frequency current acts as an excitatory agent and results in muscle contraction. Therefore, this technique cannot be used to treat unwanted motor activities.

Electrical stimulation with medium-frequency alternating electrical currents (MFAEC; 2-50 kHz) can inhibit peripheral motor nerve activities and force production, when implanted directly on top of the peripheral nerve of interest. However, this strategy is rather invasive. Thus, the administration of transcutaneous medium-frequency alternating electrical currents (tMFAEC), i.e. administration of electrical currents through the skin, might offer a solution. However, the effects of tMFAEC on motor nerve inhibition remains largely unknown. Theoretically, the administration of tMFAEC on the sensory nerve may even result in partial or complete (reversible) nerve block thereby serving as an anesthesia in order to perform surgical or painful procedures.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE

Patients suffering from neurological disorders often experience undesired sensorimotor activities e.g. hypersensitisation, spasticity and hyper- and dystonia. To overcome these disabilities, various therapeutic interventions e.g. oral medications, botulinum neurotoxin injections, local anaesthetics, transcutaneous electrical stimulation and surgeries are implemented. However, these often do not offer permanent solutions. Electrical stimulation with medium-frequency alternating electrical currents (MFAEC; 2-50 kHz) can inhibit peripheral motor nerve activities and force production, when implanted directly on top of the peripheral nerve of interest. The administration of transcutaneous medium-frequency alternating electrical currents (tMFAEC), i.e. administration of electrical currents through the skin, might offer a less-invasive alternative. Theoretically, the administration of tMFAEC on the sensory nerve may even result in partial or complete (reversible) nerve block thereby serving as an anesthesia in order to perform surgical or painful procedures. A promising pre-clinical study of Kim et al.1 already demonstrated that tMFAEC stimulation at 10 kHz can partially inhibit both sensory perception and motor activity.

1. AIM AND HYPOTHESIS

   The primary aim of this study is to confirm the previous results in literature.

   It is hypothesized that tMFAEC stimulation on the distal median nerve would:
   * Reduce sensory perception in the index and middle fingers
   * Inhibit force production by the index and middle fingers
2. OUTCOME MEASURES 2.1 Primary outcome measure

   Assessment of peripheral sensory perception and force production in the index and middle finger when tMFAEC is applied with a fixed current intensity of 31.5mA at a frequency of 10kHz to the distal median nerve. The peripheral sensory perception will be measured with the Semmes-Weinstein monofilament examination and pressure algometry that measures tactile and pressure sensation, respectively. The assessment of force production will be measured with an electronic handheld dynamometer (CompuFet 2).

   2.2 Secondary outcome measures I. Confirmation of participant's safety of tMFAEC by determining the maximum capacity tolerable for a participant. Determination is assessed by gradually increasing the tMFAEC to individual pain threshold with a maximum current intensity of 35mA.

   II. Evaluation of the effect of a different frequency i.e. 2kHz with a fixed current intensity of 31.5mA on the level of sensorimotor inhibition.

   III. Evaluation of the effect of two substantially different electrodes (i.e. PALS Platinum Electrodes 50x50mm and 3M™ Red Dot™ Elektrode foam basis klevende gel, 2228) on the level of sensorimotor inhibition.

   IV. Evaluation of the level of impedance in relation with frequency and the effect of impedance on the level of sensorimotor inhibition.

   V. Evaluation of effect of the depth of the median nerve at mid-forearm level on the level of sensorimotor inhibition.
3. STUDY PROCEDURE AND MEASUREMENTS

First, the location and depth (in mm) of the median nerve will be identified using a Sono Site Xporte ultrasound machine with a high-frequency linear transducer HFL38 (15-6MHz). The skin over the median nerve will be cleaned with ether. Electrode 1 will be placed on the skin overlying the median nerve near the transverse carpal ligament. Electrode 2 will be placed 7 cm superior to electrode 1, right above the course of the median nerve in the forearm (identified with ultrasound). Electrode placement will be slightly adjusted if MFAC stimulation induced undesired muscle contraction secondary to direct stimulation of the neuromuscular junction or asynchronous firing of the nerve. For example, if stimulation will cause thenar muscle contraction, the location of the electrodes will be moved slightly (approximately 0.5 cm) toward the ulnar or the proximal side.

Subsequently, the participants will be seated on a chair and their arms will be positioned on a testing table. The height of the chair will be adjusted such that participants can put their arms on the table with both shoulders at approximately 35° of abduction and 45° of flexion and elbows at approximately 45° of flexion. A rigid Styrofoam™ board will be used to support both wrists and forearms.

To apply tMFAEC stimulation through surface electrodes (PALS Platinum Electrodes 50x50mm and 3M™ Red Dot™ Elektrode foam basis klevende gel, 2228) and to measure the level of impedance, we will use the following device:

● DS5 Isolated Bipolar Constant Current Stimulator

In order to create a biphasic, steady, unmodulated alternating current of 10 kHz, we generate the waveform on a signal generator and deliver this to the DS5 input.

Semmes-Weinstein monofilament examination and pressure algometry:

These tests will be performed at baseline and 100% current intensity in both the 2kHz and 10 kHz stimulation group.

Tactile sensation - A set of 20 nylon monofilaments, graded according to monofilament diameter, will be used. Each monofilament will be pressed to the skin, beginning with the smallest diameter to obtain an ascending method of threshold testing. All monofilaments will be held in contact with the skin until it bends (creating a 'C-letter'), and will then be removed after 1 second. During this test, all participants will be asked to close their eyes and indicate whether or not they can sense the monofilament stimulation.

For both the 2kHz and 10 kHz, tMFAEC stimulation will be applied for 5 seconds. Then, monofilament stimulation will start 1-3 seconds after starting the tMFAEC stimulation, so that participants cannot anticipate the onset of the monofilament stimulation.

The tactile threshold will be recorded in milligram force as directed by the manufacturer and force values will be presented using a logarithmic scale.

Pressure sensation/pain - A 1 centimeter diameter algometer will be used. The pressure will be applied in a perpendicular direction using the algometer. The participants will be instructed to indicate when they feel a transition from touch/pressure to pain, corresponding to each participant's pressure pain threshold. Pressure will be increased at a rate of 1kg/cm² and released after the subject reports pain. Pressure will be applied after tMFAEC stimulation. When the pressure pain threshold is reached, tMFAEC stimulation will be stopped.

All pressure pain threshold values will be recorded in kg/cm².

Force production assessment: This test will be performed at baseline and 100% intensity.

A customised plastic frame (120 x 110 mm) with an arch will be placed underneath the palm to maintain approximately 0° wrist extension and metacarpophalangeal flexion. Next, 2 straps will be used to fix the participant's wrist and forearm to a testing platform to limit force transmission from proximal muscles and from the elbow and shoulder joints.

The participants will press a force sensor (i.e. an electronic hand held dynamometer (CompuFET 2) with the head of the proximal phalanx of each index and middle finger. The wrist and hand position will be optimised to maximise the contribution of the intrinsic hand muscles. To determine the target force, participants will be asked to press the sensors using maximum voluntary contraction (MVC). During the MVC measurements, a digital monitor will provide visual feedback on virtual finger forces, calculated as the sum of the forces produced by the index and middle fingers. The MVC measurement will be repeated 3 times and the values will be averaged.

After 3-5 practice times, the task will be repeated with MFAC stimulation. The tasks will be conducted under 4 conditions: 90-100% MVC, 100% tMFAEC stimulation at 2kHz or 10kHz and application of platinum electrodes or 3M electrodes. These 4 conditions will be repeated 3 times. Between every measurement, a 1 minute rest period will be given.

8. STATISTICAL ANALYSIS Data will be presented using the mean and standard deviation values or median and interquartile range according to the data distribution (normal or non-normal distribution, respectively).

8.1 Primary study outcome To compare the tactile threshold on the level of sensorimotor inhibition between baseline and 100% MFAC intensity (31.5mA) with two different stimulation frequencies i.e. 2kHz and 10kHz a one-way ANOVA with repeated measures (in case of a normal distribution of the data) or a Friedman test (in case no normal distribution) will be used for each of the index and middle fingers followed by a post-hoc test.

For the comparison of pressure pain thresholds among baseline and 100% intensity of tMFAEC stimulation in the index and middle fingers and to compare finger forces between the three phases using normalized mean and minimum values, a one-way ANOVA with repeated measures or a Friedman test will be used. To evaluate the exact significant differences, a Student t test or the Wilcoxon signed-rank test with a Bonferroni adjustment will be used.

The level of significance will be set at p < 0.05.

8.2 Secondary study outcomes Confirmation of participant's safety of tMFAEC by determining the maximum current intensity capable to a participant will be presented with descriptive statistics.

Evaluation of the effect of two different electrodes with substantially different materials on the level of sensorimotor inhibition will be presented with descriptive statistics.

8.3 Interim analysis N.A.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers > 18 years old

Exclusion Criteria:

* Musculoskeletal pain
* Neurologic disorder
* Diabetes mellitus
* Hypertension
* Autoimmune disease
* Any type of surgical history
* Allergy for the electrode patches

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Sensory perception: tactile sensation | 10 minutes
  Assessment of tactile sensory perception in the index finger when tMFAEC is applied with a fixed current intensity of 31.5mA at a frequency of 10kHz to the distal median nerve. The tactile sensory perception will be measured with the Semmes-Weinstein monofilament examination. Tactile sensation will be measured in grams (g).
Force Production | 5 minutes
  Assessment of force production in the index and middle finger when tMFAEC is applied with a fixed current intensity of 31.5mA at a frequency of 10kHz to the distal median nerve. The assessment of force production will be measured with an electronic handheld dynamometer (MicroFET2) and the peak force will be measured in Newton (N).
Sensory perception: pressure sensation | 5 minutes
  Assessment of pressure sensory perception in the index finger when tMFAEC is applied with a fixed current intensity of 31.5mA at a frequency of 10kHz to the distal median nerve. The pressure sensory perception will be measured with a pressure algometer. Tactile sensation will be measured in kilograms per squared centimeter (kg/cm²).

SECONDARY OUTCOMES:
Safety: peak current intensity | 2 minutes
  Confirmation of participant's safety of tMFAEC by determining the maximum capacity tolerable for a participant. Determination is assessed by gradually increasing the tMFAEC to individual pain threshold with a maximum current intensity of 35mA.
Effect of different frequency | 20 minutes
  Evaluation of the effect of a different frequency i.e. 2kHz with a fixed current intensity of 31.5mA on the level of sensorimotor inhibition. Sensory perception tests and force production assessment will be performed as described in the primary outcomes.
Effect of different type of electrode | 20 minutes
  Evaluation of the effect of two substantially different electrodes (i.e. PALS Platinum Electrodes 50x50mm and 3M™ Red Dot™ Elektrode foam basis klevende gel, 2228) on the level of sensorimotor inhibition. Sensory perception tests and force production assessment will be performed as described in the primary outcomes for both electrodes.
Effect of the depth of the median nerve | 2 minutes
  Evaluation of effect of the depth of the median nerve at mid-forearm level will be measured. The depth will be measured with the Sonosite X-porte Ultrasound machine and will be measured in millimeters (mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology, Hasselt, Belgium

REFERENCES:
- [Derived] Maris S, Brands M, Lenskens D, Braeken G, Kemnitz S, Vanhove H, Mc Laughlin M, Meesen R, Brone B, Stessel B. Transcutaneous electrical nerve inhibition using medium frequency alternating current. Sci Rep. 2022 Sep 1;12(1):14911. doi: 10.1038/s41598-022-18974-3. PMID 36050354